CLINICAL TRIAL: NCT02372201
Title: Effects of Fasting and Hydro Colon Therapy Plus Probiotics on Abundance and Diversity of GI Microbiota in Intolerances and Irritable Bowel Syndrome
Brief Title: Effects of Fasting and Hydro Colon Therapy Plus Probiotics on GI Microbiota in Intolerances and Irritable Bowel Syndrome
Acronym: MicFFGAH2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Univ. Doz. Dr. Alexander Haslberger, Univ. Dozent, University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MicrobColonIrrFFG2013
Record Dates: First submitted 2015-01-12; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Irritable Bowel Disease
Keywords: irritable bowel disease; microbiota; hydro colon therapy; food intolerance
MeSH Terms: conditions — Irritable Bowel Syndrome; Food Intolerance | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydro Colon Therapy plus probiotic (Experimental): Hydro Colon therapy including 2-5 washes in 3 weeks, probiotic intervention for 5 weeks after end of hydro Colon therapy
  Interventions: Other: Hydro Colon Therapy plus probiotic

INTERVENTIONS:
Other: Hydro Colon Therapy plus probiotic — Probiotic intervention was done after 2-5 cycles of hydro colon therapy.

SUMMARY:
Consequences of Colon Hydrotherapy plus probiotic intervention on composition of GI microbiota and well being are analysed in subjects claiming GI inconveniences due to Irritable Bowel Syndrome or food intolerances.

DETAILED DESCRIPTION:
Study objectives: Analysis of consequences of Hydro Colon Therapy plus probiotic intervention on GI microbiota and well being.

Study group: 78 subjects, inclusion criteria: 20-50yrs; under consultation at doctors or nutritionists because of claimed food inconveniences or Irritable Bowel Syndrome. exclusion criteria: antibiotics treatment and specified complex diseases.

Intervention: Hydro colon therapy 2- 5 washes within 3 weeks. probiotic intervention after end of Hydro colon therapy for 6 weeks ( DUOLAC® bacterial strains per capsule: Lactobacillus plantarum, Streptococcus thermophiles, Lactobacillus acidophilus, Lactobacillus rhamnosus, Bifidobacterium lactis, Bifidobacterium longum, and Bifidobacterium breve, fructooligosaccharides, 200 µg folic acid, 2.50 µg vitamin B12 and 55 µg selenium (all amounts corresponding to 100% of daily requirement). Control group: Vitamin B complex: 10µg cobalamin, 450µg folic acid, and 55 µg selenium.

Sample collection: standardized Feces collection, T1, before colon hydrotherapy, T2, immediately after colon hydrotherapy 2-5 washes of fasting ; T3, after six weeks of probiotic or Control intervention Analysis: standardizes food frequency questionnaire before and after intervention.

Feces analysis based on 16 S ribosomal DNA (rDNA) PCR DGGE and quantitative PCR (qPCR) and bioinformatic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects under consultation at doctors or nutritionists for Inflammatory Bowel Syndrome (IBD) of food intolerances

Exclusion Criteria:

* Pregnancy
* Antibiotic therapy 0,5 yrs before start
* Hormone therapies
* Malignant diseases
* Subjects were asked to avoid dietary supplements 4 weeks before and during the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
microbiota structure, using 16 S ribosomal based gradient electrophoresis ( DGGE) | 7- 8 weeks hydro colon washes plus probiotic
  Microbiota were analysed for abundance of main microbiota groups and microbiota diversity using 16 S ribosomal based gradient electrophoresis ( DGGE). Abundance is shown in DNA copies/g feces; diversity as number of bands/ sample and by bioinformatic analysis
Gastrointestinal comfort, measured by Visual Analog Scale | 7- 8 weeks hydro colon washes plus probiotic
  Gastrointestinal comfort was analysed by a standardised questionnaire. Pain was measured by Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Haslberger, Principal Investigator — UNIVIE
Locations (1):
- Dep. for Nutritional Sciences, University of Vienna, Vienna, Select Your State, Austria